CLINICAL TRIAL: NCT00368576
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group, Repeat Dose Study to Assess the Effect of SB-480848 on Overall Asthma Control in Adult Subjects With Persistent Asthma Controlled on Stable, Low-dose, Inhaled Corticosteroids
Brief Title: A Study To Determine The Effect Of SB-480848 On Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: LPL107629
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Atherosclerosis
Keywords: SB-480848; methacholine challenge; asthma; inhaled steroid
MeSH Terms: conditions — Atherosclerosis; Asthma | interventions — darapladib; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB 480848, tablets
  Other Names: SB 480848; tablets

SUMMARY:
The purpose of this study is to compare the effects of SB-480848 with placebo in subjects with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects who have documented persistent asthma for at least 3 months
* Subjects must have been on a stable, low-dose ICS for a minimum of 4 weeks prior to the screening visit.
* Aged 18-65 years, at screening
* FEV1 greater than or equal to 70% predicted (ECCS, 1993)
* Subjects must show an increase in FEV1 greater than or equal to 12% (and an absolute change >200mL) within 30 minutes following inhalation of 4 puffs of albuterol/salbutamol or 1 nebulized treatment of 2.5mg or have historical, documented evidence of reversibility, within 12 months prior to screening
* Subjects must be willing to replace their inhaled, short-acting β2-agonist with study provided albuterol/salbutamol
* Patient must be capable of giving informed consent and comply with the study requirements and timetable.

Inclusion Criteria following run in period (Prior to randomisation) Subjects will be screened based on the inclusion and exclusion criteria noted above.

During the run-in period [Day -14 to Day 1], subjects will be asked to maintain a diary card and document the number of puffs of rescue inhaled, short-acting β2-agonists taken, asthma-related symptoms and night time awakenings as well as morning and evening PEF measurements.

On the morning of Day 0, subjects will be eligible for randomisation into the study if all of the following criteria are met:

* Subjects required, on average less than or 2 puffs per day of study provided albuterol/ salbutamol during the last 7-day period prior to Day 0 [from Day -7 to Day 1]
* Subjects had asthma symptoms on less than or 5 out of the last 7 consecutive days of the run-in period
* FEV1 greater than or equal to 70% predicted (ECCS, 1993).
* FEV1 must be within ± 15% of the FEV1 value at beginning of screening.
* Compliance with completion of the diary card.

Exclusion criteria:

* The patient has life threatening asthma. A research patient must not have been hospitalized two or more times in the last year prior to Day 0 due to asthma and must not have been hospitalized within 6 months prior to Day 0
* Subjects with daily asthma-related symptoms.
* Subjects taking any of the medications listed in the protocol for the listed interval prior to the screening visit or during the study:
* Subjects with historical or current evidence of any other disease.
* Subjects with clinically significant abnormal findings on physical exam or other screening procedures.
* Subjects who have received an investigational product within 30 days or 5 half-lives [whichever is longer] prior to the first dose of study medication
* Subjects who have tested positive for hepatitis C antibody, hepatitis B surface antigen or HIV.
* Subjects with history of drug or alcohol abuse
* Positive drug (not related to known medications the subject is taking at time of screening), alcohol or cotinine/carbon monoxide (CO) test at screening or at Day 0
* Subjects with a history of regularly drinking more than 2 (females)/3 (males) units of alcohol a day.
* Pregnant or nursing female subjects.
* Female subjects of childbearing potential with an unwillingness to agree to one of the methods of contraception listed in the protocol.
* Subjects who suffer from any medical condition which in the opinion of the investigator would compromise patient safety or ability to comply with study procedures
* Subjects who are current smokers or have given up smoking within the previous six months or who have a smoking history > 10 pack years.
* Subjects with history of an upper or lower respiratory tract infection or symptoms (including the common cold) within 2 weeks prior to first dose of study medication
* Subjects who have donated more than 500ml of blood within 56 days prior to the first dose of study medication
* Subjects who are currently receiving potent 3A4 inhibitors be excluded.
* Subjects on β-adrenergic receptor blockers within 3 months prior to screening visit
* Subjects previously hospitalized as a result of a methacholine challenge

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
FEV1 | 6 hours post-dose, Days 7, 14 and 21

SECONDARY OUTCOMES:
Methacholine challenge Amounts of certain chemicals/proteins in blood Amount of drug in the blood | before dosing and after 21 days of dosing
Measurements of FEV1 following single doses of SB-480848 and placebo.
Measurements of PC20 on Day 21 +24hrs after dosing with SB-480848 and placebo. | Day 21 +24hrs after dosing
Blood drug levels of SB-553253 [metabolite of SB-480848] may be assessed, as appropriate.
Urinary leukotriene concentrations after 21 days of dosing with SB-480848 and Placebo. | after 21 days
Blood levels of LpPLA2 and CD62 concentrations over 21-day dosing period with SB-480848 and placebo | over 21-day dosing period
Measurements of FEF25-75 and peak expiratory flow following single and repeat oral doses of SB-480848.
Assessment of vitals, ECGs, safety labs and number of puffs of rescue inhaled, short-acting β2-agonists taken, asthma-related symptoms and night time awakenings, number of subjects withdrawn due to worsening of asthma on SB- 480848 and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (4):
  - GSK Investigational Site, Cypress, California
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Spartanburg, South Carolina
- Germany (3):
  - GSK Investigational Site, Neu-Ulm, Bavaria
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: LPL107629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LPL107629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LPL107629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LPL107629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LPL107629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LPL107629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LPL107629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register